CLINICAL TRIAL: NCT03042767
Title: Anti-LPS Antibody in Pediatric Nonalcoholic Fatty Liver Disease
Brief Title: Anti-LPS Antibody Treatment for Pediatric NAFLD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Miriam Vos, MD (Other)
Collaborators: Advanced MR Analytics AB (Industry); Immuron Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Miriam Vos, MD, Associate Professor, Emory University
Organization: Emory University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00084686
Record Dates: First submitted 2017-02-02; First posted 2017-02-03 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-04

CONDITIONS: Nonalcoholic Fatty Liver Disease (NAFLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IMM-124E Group (Experimental): Participants with nonalcoholic fatty liver disease (NAFLD) will receive 600mg of IMM-124E powder three times daily for twelve weeks.
  Interventions: Biological: IMM-124E
- Placebo Group (Placebo Comparator): Participants with nonalcoholic fatty liver disease (NAFLD) will receive placebo powder three times daily for twelve weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: IMM-124E — IMM-124E is a hyper-immune, bovine colostrum (milk) powder with flavoring.
  Arms: IMM-124E Group
Other: Placebo — Matched Placebo
  Arms: Placebo Group

SUMMARY:
The main objective of this pilot study is to evaluate whether 12 weeks of IMM-124E in children with nonalcoholic fatty liver disease (NAFLD) in combination with standard of care treatment will decrease inflammation in the liver as measured by alanine transaminase (ALT). Specifically, investigators will measure percent change in ALT from Week 0 to Week 12 in treatment compared to placebo.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo controlled, three month treatment trial of children aged 6-19 years. Participants will be recruited from the Children's Healthcare of Atlanta pediatric liver clinical practice.The purpose of this study is to evaluate if a three month treatment with IMM-124E (a bovine colostrum enriched with anti-LPS antibodies) in combination with standard of care lifestyle advice is safe and leads to greater improvement in hepatic inflammation, insulin sensitivity, and blood lipids in children with nonalcoholic fatty liver disease (NAFLD) compared to placebo with standard of care treatment. Investigators also seek to define the mechanism of action in response to three months of treatment with IMM-124E.

ELIGIBILITY:
Inclusion Criteria:

* Nonalcoholic fatty liver disease (NAFLD) diagnosis confirmed by liver biopsy or MRI
* ALT ≥ 2 x ULN at screening (girls ≥ 46, boys ≥ 54)
* Written informed parent consent and child assent
* Willingness to take IMM-124E or placebo powder 3 x daily for 12 weeks
* At least 2 months of attempted lifestyle changes after diagnosis

Exclusion Criteria:

* Disease or condition deemed by physician to interfere with absorption, digestion, or mechanism of intervention of drug
* Diagnosis of diabetes and an HbA1c of > 9%
* Change in supplement or anti-oxidant therapy within past 90 days (must be on a stable dose and willing to continue it throughout the trial or not on any vitamin or supplement, includes SAMe, vitamin E, betaine, Milk thistle etc)
* Use of probiotics or antibiotics in the past 30 days
* Use of anti-NAFLD medications (metformin, thiazolidinediones, UDCA) in the 30 days prior to randomization
* Acute illness within past 2 weeks prior to enrollment (defined as fever > 100.4ºF)
* Planned pregnancy, nursing an infant, confirmed or suspected to be pregnant between screening and time of study enrollment
* Evidence of other chronic liver disease other than NAFLD (Hepatitis B and C, Alpha-1 antitrypsin, Wilson's disease)
* Intolerance to lactose or dairy-based products
* Unable to have blood drawn at study visits
* Unwillingness to provide and/or collect stool samples
* Current gastrointestinal (GI) bleeding or inflammatory bowel disease (irritable bowel disease (IBD), colitis)
* Current enrollment in another therapeutic clinical trial or receipt of an investigational study drug within 6 months prior to study enrollment
* Participants who are not able or willing to comply with the protocol or have any other condition that would impede compliance or hinder completion of the study, in the opinion of the investigator

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Vos, MD, MSPH, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 40 participants were enrolled, 15 of them screenfailed. 25 participants were randomized.
Period: Overall Study
Arm/Group | IMM-124E Group | Placebo Group
Started | 12 | 13
Completed | 11 | 11
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IMM-124E Group | Placebo Group | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 13 | 25
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 7 | 17
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Alanine Aminotransferase (ALT) Level
Description: Percent change in ALT level from baseline to end of treatment.
Time Frame: Baseline (Week 0), End of Treatment (Week 12)
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | IMM-124E Group | Placebo Group
Number analyzed (Participants) | 11 | 11
percentage change | 11.99 (25.87) | -7.99 (16.54)

2. Secondary Outcome: Percent Change in Fasting Glucose Level
Description: Fasting glucose level will be collected via blood draw. Percent Change in glucose levels between baseline and end of treatment.
Time Frame: Baseline (Week 0), End of Treatment (Week 12)
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | IMM-124E Group | Placebo Group
Number analyzed (Participants) | 11 | 11
percentage change | 4.55 [-1.14 to 16.05] | 1.11 [-6.54 to 3.49]

3. Secondary Outcome: Change in Fasting Insulin Level
Description: Fasting insulin level will be collected via blood draw. Change is the difference in insulin level from baseline to end of treatment.
Time Frame: Baseline (Week 0), End of Treatment (Week 12)
Population: Data were not analyzed due to funding limitation.
Arm/Group | IMM-124E Group | Placebo Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Hemoglobin A1C Level
Description: Hemoglobin A1C Level will be collected via blood draw. Change is the difference in hemoglobin AIC level from baseline to end of treatment.
Time Frame: Baseline (Week 0), End of Treatment (Week 12)
Population: Data were not collected. Hemoglobin A1c was only used as a screening lab, it was not measured throughout the study - change cannot be measured
Arm/Group | IMM-124E Group | Placebo Group
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Adipose Tissue Insulin Resistance (Adipo-IR)
Description: Adipo-IR will be collected via blood draw. It is calculated as fasting non-esterified fatty acids x fasting insulin.
Time Frame: Baseline (Week 0), End of Treatment (Week 12)
Population: Data were not analyzed due to funding limitation.
Arm/Group | IMM-124E Group | Placebo Group
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Triglyceride/HDL (TG/HDL) Ratio
Description: The TG/HDL ratio is the proportion of triglyceride levels in relation to HDL (good cholesterol). Change is defined as the difference in the TG/HDL ratio from baseline to the end of treatment.
Time Frame: Baseline (Week 0), End of Treatment (Week 12)
Population: Data were not analyzed due to funding limitation.
Arm/Group | IMM-124E Group | Placebo Group
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percent Change in Blood Glucose Level
Description: The blood glucose level will be monitored via an oral glucose tolerance test (OGTT) at baseline and at the end of treatment. During the OGTT, the glucose level will be tested by a blood draw every thirty minutes for two hours. Percentage change between glucose measurements taken at baseline and at the end of treatment is reported.
Time Frame: Baseline (Week 0), End of Treatment (Week 12)
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | IMM-124E Group | Placebo Group
Number analyzed (Participants) | 11 | 11
percentage change | 2.11 [-3.06 to 16.05] | 1.16 [-6.54 to 3.49]

8. Secondary Outcome: Change in Insulin Levels
Description: The insulin level will be monitored via an oral glucose tolerance test (OGTT) at baseline and at the end of treatment. During the OGTT, the insulin level will be tested by a blood draw every thirty minutes for two hours. Change is described as the difference between insulin measurements taken at baseline and at the end of treatment.
Time Frame: Baseline (Week 0), End of Treatment (Week 12)
Population: Data were not analyzed due to funding limitation.
Arm/Group | IMM-124E Group | Placebo Group
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Percent Change in Body Mass Index (BMI) Z-Score
Description: BMI will be calculated from height and weight and converted into a z-score. Body mass index z-scores are measures of relative weight adjusted for age and sex.Change is the difference in BMI z-scores from base line to end of treatment.
Time Frame: Baseline (Week 0), End of Treatment (Week 12)
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | IMM-124E Group | Placebo Group
Number analyzed (Participants) | 11 | 11
percentage change | 1.66 [-0.46 to 2.38] | -0.48 [-3.77 to 2.83]

10. Secondary Outcome: Percent Change in Visceral Adiposity
Description: Visceral adiposity will be measured with a magnetic resonance imaging (MRI) scan. Visceral adipose tissue is a hormonally active component of total body fat.
Time Frame: Baseline (Week 0), End of Treatment (Week 12)
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | IMM-124E Group | Placebo Group
Number analyzed (Participants) | 11 | 11
percentage change | 1.23 (8.63) | 1.77 (9.07)

11. Secondary Outcome: Percent Change in Hepatic Fat Percent
Description: Hepatic fat percent will be measured with a magnetic resonance imaging (MRI) scan. Hepatic fat percent is the percentage of fat within the liver.
Time Frame: Baseline (Week 0), End of Treatment (Week 12)
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | IMM-124E Group | Placebo Group
Number analyzed (Participants) | 11 | 11
percentage change | -5.70 (16.80) | -6.61 (17.15)

12. Secondary Outcome: Percent Change in Waist Circumference
Description: Waist circumference will be measured in centimeters using measuring tape.
Time Frame: Baseline (Week 0), End of Treatment (Week 12)
Measure: Median (Inter-Quartile Range); unit: percentage change
Arm/Group | IMM-124E Group | Placebo Group
Number analyzed (Participants) | 11 | 11
percentage change | 2.29 [-0.88 to 4.29] | 0.76 [-0.33 to 1.50]

13. Secondary Outcome: Percent Change in PROMIS Fatigue Questionnaire Score
Description: The PROMIS Fatigue questionnaire evaluates a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Fatigue is divided into the experience of fatigue (frequency, duration, and intensity) and the impact of fatigue on physical, mental, and social activities. It assesses fatigue over the past seven days. A higher score represents more symptoms of fatigue.
Time Frame: Baseline (Week 0), End of Treatment (Week 12)
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | IMM-124E Group | Placebo Group
Number analyzed (Participants) | 11 | 11
percentage change | -10.17 (14.90) | -4.67 (17.18)

14. Secondary Outcome: Percent Change in PROMIS Depression Questionnaire Score
Description: The PROMIS Depression instruments assess self-reported negative mood (sadness, guilt), views of self (selfcriticism, worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose). It assesses depression over the past seven days. A higher score represents more symptoms of depression.
Time Frame: Baseline (Week 0), End of Treatment (Week 12)
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | IMM-124E Group | Placebo Group
Number analyzed (Participants) | 11 | 11
percentage change | -7.68 (17.00) | 3.62 (11.97)

15. Secondary Outcome: Percent Change in PROMIS Anxiety Questionnaire Score
Description: The PROMIS Anxiety instruments measure self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness). Anxiety is best differentiated by symptoms that reflect autonomic arousal and experience of threat. Each assesses anxiety over the past seven days. A higher score represents more symptoms of anxiety.
Time Frame: Baseline (Week 0), End of Treatment (Week 12)
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | IMM-124E Group | Placebo Group
Number analyzed (Participants) | 11 | 11
percentage change | -13.78 (16.39) | -4.89 (13.89)

16. Secondary Outcome: Composite Metabolic Improvement
Description: Composite metabolic improvement is defined as greater than 10% improvement in TG/HDL ratio, improvement in insulin resistance, and greater than 10% improvement in ALT.
Time Frame: End of Treatment (Week 12)
Population: Data were not analyzed due to funding limitation.
Arm/Group | IMM-124E Group | Placebo Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | IMM-124E Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 8/12 | 10/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMM-124E Group (N=12) | Placebo Group (N=13)
Abdominal pain (General disorders) | 1 (1) | 2 (2)
Abnormal glucose result (Endocrine disorders) | 2 (3) | 5 (8)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomit (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Headache (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT03042767/Prot_SAP_000.pdf